CLINICAL TRIAL: NCT00331370
Title: Hypertension Related Damage to the Microcirculation in South Asian: Emergence,Predictive Power and Reversibility
Brief Title: Hypertension Related Damage to the Microcirculation in South Asian: Emergence, Predictive Power and Reversibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Imperial College London (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: DHCPP00493
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2006-05-31 (Estimated); Status verified 2006-05

CONDITIONS: Hypertension; Diabetes; Cardiovascular Disease; Retinopathy
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Cardiovascular Diseases; Retinal Diseases

INTERVENTIONS:
Behavioral: GP training and Health Education

SUMMARY:
Damage to very small blood vessels is a consequence, but can also precede high blood pressure. Such damage, measured by disturbances in the vessels in the retina (back of the eye) is a strong predictor of heart disease and stroke. South Asian people have one of the highest rates of hypertension in the world (30% in adults). In Pakistan, this is usually severe, undetected and untreated. The Wellcome Trust has already funded a study of blood pressure control in adults and children in this population. We propose a substudy, taking photographs of the retina and making measurements of the vessels, to determine whether such blood pressure related changes occur at an early age in young children with a family history of high blood pressure compared to those without, whether such changes predict an increase in blood pressure over time, and whether, in adults, such changes can be reversed by blood pressure treatment. The hypothesis of our study is: young offspring of South Asian people with hypertension have a disturbed microcirculation, as assessed by abnormalities of retinal vessels, compared to offspring of normotensive parents. Our 2nd hypothesis is: Abnormal retinal vascular geometry will improve proportionately to achieved reductions in BP.

DETAILED DESCRIPTION:
Background

The role of the microcirculation is increasingly being recognized in the etiopathogenesis of cardiovascular disease. Delays in this recognition are in part due to the difficulty of studying the microcirculation non-invasively, in large numbers of individuals. Retinal vessels provide an easily accessible "window" to the microcirculation. Abnormalities of the retinal vasculature have been shown to be associated with cardiovascular risk factors and all cause mortality. Non-invasive assessment of the retinal circulation presents a valuable opportunity to study the structure and function of the microvasculature

Aims of the project

To compare geometry of retinal microvasculature of 1) hypertensive vs normotensive adults, 2) children aged 10 to 14 years of hypertensive parent (test group) versus normotensive parent (control group), and, 3) to assess the impact of blood pressure lowering on these changes over 2 years.

Primary outcome would be abnormal retinal geometry defined as the composite outcome of a) abnormal arteriolar length: diameter ratios (a measure of relative arteriolar narrowing), b) narrowed branching angles (an indicator of arteriolar rarefaction), or c) disturbed junction exponents (a marker of endothelial dysfunction.

Significance of the study

If successful, this work could be extended to address future questions, including the predictive value of these abnormalities for development of diabetes and hypertension as well as CVD; to explore further the role of microvascular disturbances in disease etiology, and to assess the impact of drug therapy on these abnormalities and their relationship to outcomes in the South Asian population

ELIGIBILITY:
Inclusion Criteria:

All subjects aged 9 years or over residing in randomly selected communities

Exclusion Criteria:

Pregnancy

Those who have severe co-morbid conditions

Patients with known history of glaucoma will be excluded from our study because instillation of mydriatic drops was thought to be hazardous for them.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2880
Dates: Start 2006-05; Study Completion 2009-06

PRIMARY OUTCOMES:
Primary outcome would be abnormal retinal geometry defined as the composite outcome of a) abnormal arteriolar length: diameter, b) narrowed branching angles, or c) disturbed junction exponents.

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD, MPH, Principal Investigator — Aga Khan University; Nish Chaturvedi, MD, MFPHM, Study Chair — Imperial College London; Alun Hughes, MD, Phd, Study Chair — Imperial College London; Juanita Hatcher, Phd, MSc, Study Chair — Aga Khan University; Simon Thom, MD, FRCP, Study Chair — Imperial College London; Khabir Ahmad, MD, MSc, Study Chair — Aga Khan University; Muhammad Saleem Khan, MSc Epi&Bio, Study Chair — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan